CLINICAL TRIAL: NCT02150850
Title: Quebec Registry for Atypical Femur Fractures
Status: Recruiting | Type: Observational
Sponsor: McGill University (Other)
Collaborators: Fonds de la Recherche en Santé du Québec (Other Government); McGill University Health Centre/Research Institute of the McGill University Health Centre (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Dr. Suzanne Morin, Associate Professor, McGill University
Other Study IDs: A00-M23-12A
Record Dates: First submitted 2014-05-20; First posted 2014-05-30 (Estimated); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Atypical Femur Fracture
Keywords: Femoral Fractures; Subtrochanteric Fractures; Osteoporotic Fractures; Fractures, Spontaneous; Stress Fractures; Bone Fractures; Hip Fractures; Osteoporosis
MeSH Terms: conditions — Femoral Fractures; Hip Fractures; Osteoporotic Fractures; Fractures, Spontaneous; Fractures, Stress; Fractures, Bone; Osteoporosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — AFF patients only will be asked to deposit 2 ml of saliva into a collection tube using a standardized protocol. Individuals unable to produce 2ml of saliva will be asked to perform at least two buccal swabs.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Registry: Patients who have who have sustained an AFF that consent to participating in the registry only.
- Cases: Patients who have sustained an AFF that consent to participating in the registry and undergoing EOS® imaging.
- Controls: For each case we will identify one age- (± 5 years), sex-, height- (± 6 cm) and cumulative bisphosphonate or denosumab exposure ( ±2 years) matched control who has not sustained an AFF to undergo EOS® imaging.

SUMMARY:
Bisphosphonates are recommended as first-line agents to reduce fracture risk in patients with osteoporosis and have in general an excellent safety profile. However, recent reports have noted that prolonged use of bisphosphonates may be associated with rare but serious adverse effects, namely atypical femur fractures (AFF), an atraumatic subset of subtrochanteric and diaphyseal fractures.

The overarching aim of this project is to contribute to the characterization of clinical, biomechanical, radiological and genetic predictors of AFF, associated or not with bisphosphonate and-or denosumab therapy. AFF arise on the lateral (external) aspect of the subtrochanteric and diaphyseal regions of the femur, regions subjected to high mechanical loads. Because of this unique distribution, the investigators hypothesis is that patients with AFF demonstrate specific geometrical variations of their femur whereby baseline tensile forces applied to the lateral cortex are higher and might favour the appearance of these rare stress fractures. Measurements to investigate these geometric variations with be calculated from 3D images reconstructed using scans procured using the EOS® low irradiation 2D-3D X-Ray scanner.

ELIGIBILITY:
Inclusion Criteria:

* age 45 years and older
* men and women from Quebec who sustain (or have sustained) an AFF (complete or incomplete), as defined by the American Society of Bone and mineral Research (ASBMR) International Task Force on AFFs (Shane E et al J Bone Miner Res 2014;29:1-24)

Exclusion Criteria:

* inability to consent
* disorders of bone metabolism other than osteoporosis
* active cancer
* life expectancy less than 12 months.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have sustained an AFF.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2012-04; Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Predictors associated with AFFs | Baseline
  Measured as the frequency of possible risk factors including demographic and clinical characteristics.

SECONDARY OUTCOMES:
Differences in lower limb geometric parameters between cases and controls | Baseline
  Measured from 3D images reconstructed using scans procured using the EOS® low irradiation 2D-3D X-Ray scanner.

OTHER OUTCOMES:
Change from baseline in functional impairment | 6- 12- 24- 36- months post fracture
  Measured using the Lower Extremity Functional Scale (LEFS).
Change in global function status | 6- 12- 24- 36- months post fracture
  Measured using The Reintegration to Normal Living Index (RNLI).

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Morin, MD MSc, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- Montreal General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No